CLINICAL TRIAL: NCT02230748
Title: Left-Atrium-Appendage Occluder Register - GErmany
Acronym: LAARGE
Status: Completed | Type: Observational
Sponsor: Stiftung Institut fuer Herzinfarktforschung (Other)
Responsible Party: Sponsor
Other Study IDs: LAARGE
Record Dates: First submitted 2014-08-29; First posted 2014-09-03 (Estimated); Last update posted 2018-09-06 (Actual); Status verified 2018-09

CONDITIONS: Atrial Fibrillation; Stroke
Keywords: LAA; LAA-Occluder; Atrial Fibrillation; AF
MeSH Terms: conditions — Atrial Fibrillation; Stroke

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
* Evaluation of safety and effectiveness of implantable LAA occluder in clinical practice
* Indication: For which reasons is the indication for implantation of LAA-Occluder put for patients with atrial fibrillation?
* Safety: How save is the implantation of LAA-Occluders?
* Effectiveness: How effective is implantation of LAA-Occluders in daily clinical practice?
* Concomitant treatment: Which concomitant treatment is prescribed for patients with LAA-Occluder?

DETAILED DESCRIPTION:
LAARGE aims to show the care reality of patients whose left atrial appendage (LAA) is closed by an implantable medical device. In particular the following questions should be answered:

* Indication: For which reasons is the indication for implantation of LAA-Occluder put for patients with atrial fibrillation?
* Safety: How save is the implantation of LAA-Occluders (procedural, in hospital and in the long term course)? How frequent are bleeding complications and what is the relation of observed and expected bleeding complications (according HAS-BLED score)?
* Effectiveness: How effective is implantation of LAA-Occluders in daily clinical practice (in hospital and in the long term course)? How frequent are strokes and what is the relation of observed and expected strokes (according CHADS-VASC score)?
* Concomitant treatment: Which concomitant treatment is prescribed for patients with LAA-Occluder?

ELIGIBILITY:
Inclusion Criteria:

Intention to laa occluder

Exclusion Criteria:

Missing informed consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: all patients with an performed or planned LAA -Occluder
Sampling Method: Non-Probability Sample
Enrollment: 643 (Actual)
Dates: Start 2014-07; Primary Completion 2016-01 (Actual); Study Completion 2017-03-27 (Actual)

PRIMARY OUTCOMES:
Safety: clinical events with LAA occlusion | 1 year follow-up (optional 2,3,5 years)
  Documentation of reasons for LAA Occluder Implantation.
  Periprocedural and hospital: death, bleeding, pericardial effusion, reanimation, occluder dislocation and further complications.
  Long term follow-up:: death, bleeding, pericardial effusion, reanimation, occluder dislocation, further complications and patients safety.

SECONDARY OUTCOMES:
Effectiveness: LAA occlusion | 1 year follow-up (optional 2,3,5 years)
  periprocedural and hospital: Sudden or unexpected death, stroke, TIA, systemic embolism, technical success.
  Long term follow-up: Sudden or unexpected death, stroke, TIA, systemic embolism, patients satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Jochen Senges, MD, Principal Investigator — Stiftung Institut für Herzinfarktforschung (IHF)
Locations (4):
- Germany (4):
  - Klinikum Coburg, Coburg
  - Institut für Herzinfarkforschung Ludwigshafen, Ludwigshafen
  - Universitätsmedizin Mannheim, Mannheim
  - Isar Herzzentrum, München

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ansari U, Brachmann J, Lewalter T, Zeymer U, Sievert H, Ledwoch J, Geist V, Hochadel M, Schneider S, Senges J, Akin I, Fastner C. LAA occlusion is effective and safe in very high-risk atrial fibrillation patients with prior stroke: results from the multicentre German LAARGE registry. Clin Res Cardiol. 2024 Oct;113(10):1451-1462. doi: 10.1007/s00392-024-02376-8. Epub 2024 Jan 31. PMID 38294498
- [Derived] Fastner C, Brachmann J, Lewalter T, Zeymer U, Sievert H, Borggrefe M, Weiss C, Geist V, Krapivsky A, Kaunicke M, Mudra H, Hochadel M, Schneider S, Senges J, Akin I. Left atrial appendage closure in patients with a reduced left ventricular ejection fraction: results from the multicenter German LAARGE registry. Clin Res Cardiol. 2020 Nov;109(11):1333-1341. doi: 10.1007/s00392-020-01627-8. Epub 2020 Mar 31. PMID 32236717